CLINICAL TRIAL: NCT05048875
Title: Phase 2a, Randomized, Doubleblind, Placebo-controlled Trial Evaluating the Antiviral Activity, Safety and Pharmacokinetics of Repeated Oral Doses of JNJ-64281802 Against Dengue-3 Infection in a Dengue Human Challenge Model in Healthy Adults
Brief Title: An Evaluation of Repeated Oral Doses of JNJ-64281802 Against DENV-3 Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Janssen, LP (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 332; 156295 (Other: FDA IND Number); 64281802DNG2002 (Other: Janssen Protocol Number)
Record Dates: First submitted 2021-06-30; First posted 2021-09-17 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dengue
Keywords: Dengue Serotype 3; Healthy Participants
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: There are two cohorts and three groups in each cohort. Cohort 1 consists of Group 1a, Group 1b and Group 2. Cohort 2 consists of Group 3, Group 4, and Group 5. Within each group, participants will either be randomized to receive study drug or placebo.
  Four participants were enrolled in Group 1a before enrolling the remaining participants to Group 1b (12 participants) and Group 2 (14 participants) in Cohort 1. Based on the interim analysis results of Cohort 1, three groups for Cohort 2 were created. Results are posted for Cohort 1 which is complete and unblinded.
  Cohort 2 has been fully enrolled and is in progress.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subject, investigator, and clinical staff will not know which treatment group the subject has been assigned. In addition, other personnel assigned to monitor the study will not know the treatment assignment of the subject. The pharmacist will be unblinded as the study drug will be provided as bulk supplies.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - Group 1 JNJ High Dose (Experimental): Sentinel high-dose. Four participants will be enrolled in Group 1a before enrolling the remaining participants to Group 1b (12 participants total in Group 1, all same dosing regimen). Note group 1a and group 1b are combined into one arm, because the dosing regimen is the same and they were not separated during final statistical analysis.
  Interventions: Drug: Cohort 1 - Group 1 JNJ High Dose
- Cohort 1 - Group 2 JNJ Medium Dose (Experimental): Group 2 includes Medium and low dose, 14 participants total. Enrolled after completion of Group 1a.
  Interventions: Drug: Cohort 1 - Group 2 JNJ Medium Dose
- Cohort 1 - Group 2 JNJ Low Dose (Experimental): Group 2 includes Medium and low dose, 14 participants total. Enrolled after completion of Group 1a.
  Interventions: Drug: Cohort 1 - Group 2 JNJ Low Dose
- Cohort 1 - Group 1/2 Placebo (Placebo Comparator): Matching placebo. Note Group 1 placebo and group 2 placebo are combined per sponsor data analysis.
  Interventions: Drug: Cohort 1 - Group 1/2 Placebo

INTERVENTIONS:
Drug: Cohort 1 - Group 1 JNJ High Dose — High dose: 600-mg loading dose for 5 days/200-mg maintenance dose for 21 days
  Other Names: JNJ-64281802 (Sentinel high dose)
  Arms: Cohort 1 - Group 1 JNJ High Dose
Drug: Cohort 1 - Group 2 JNJ Medium Dose — Medium dose: 200-mg loading dose for 5 days/50-mg maintenance dose for 21 days
  Other Names: JNJ-64281802 (medium dose)
  Arms: Cohort 1 - Group 2 JNJ Medium Dose
Drug: Cohort 1 - Group 2 JNJ Low Dose — Low dose: 40-mg loading dose for 5 days/10-mg maintenance dose for 21 days
  Other Names: JNJ-64281802 (low dose)
  Arms: Cohort 1 - Group 2 JNJ Low Dose
Drug: Cohort 1 - Group 1/2 Placebo — Matching placebo. Note Group 1 placebo and group 2 placebo are combined per sponsor data analysis.
  Other Names: Placebo High Dose
  Arms: Cohort 1 - Group 1/2 Placebo

SUMMARY:
The investigational study drug, JNJ-64281802, is being developed for the prevention and treatment of dengue infection. This study is hypothesizing that the highest dose of the investigational study drug is superior to receiving a placebo with respect to its antiviral activity in healthy adult participants inoculated with Dengue Serotype 3.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, placebo-controlled, double-blind, interventional Phase 2a, study in normal healthy adult subjects 18 - 55 years of age, inclusive, recruited from the metropolitan Baltimore/Washington, DC area & Burlington/Vermont. The study follows an adaptive 2-stage design consisting of 2 cohorts, each with up to 3 groups. The 2 cohorts will be enrolled in a staggered manner. As a safety measure, a sentinel group of 4 participants will be enrolled in Cohort 1 (Group 1a) before enrolling the remaining participants (Group 1b and Group 2) in the cohort.

The purpose of this study is to evaluate the clinical and virologic response to repeated doses of investigation product JNJ-64281802 when administered orally in healthy, DENV and ZIKV-naïve, non-pregnant, adult volunteers who are subsequently inoculated with rDEN3delta30, a recombinant DENV-3 strain, to explore the antiviral activity of repeated oral doses of JNJ-64281802 versus placebo. The safety, tolerability, PK, and the relationship between the PK and antiviral activity of JNJ-64281802 will also be evaluated. Placebo recipients are included in the study as a control to better assess study agent associated versus non-study agent associated AEs and to act as infectivity controls following administration of rDEN3delta30.

After providing written informed consent, subjects will undergo eligibility screening, including medical history, physical examination, hematology testing, liver and renal function testing, human immunodeficiency virus (HIV) screening, hepatitis B and C screening, urinalysis, urine toxicology screening, ECG screening, alcohol breath test screening (per PI/provider discretion), COVID-19 testing (if determined necessary by the clinician or per guidelines), and serology screening for previous infection of DENV and ZIKV (Cohort 1) and DENV, ZIKV, West Nile virus, and SLEV (Cohort 2).

Serum or urine pregnancy testing will be performed on applicable persons of childbearing potential. All screening tests must be performed within 60 days of initiation of JNJ-64281802 study agent at Study Day -5 (Cohort 1) or Study Day -2 (Cohort 2). HIV screening must be performed within 2 weeks of JNJ-64281802 study agent administration. Pregnancy screening will occur at applicable screening visit(s), be repeated on the first day of JNJ-64281802 administration prior to administration, and on the day of inoculation with rDEN3delta30 prior to inoculation with rDEN3delta30. All clinically significant abnormalities will be reviewed with subjects and referral for follow-up care will be provided. Subjects will be determined to be eligible based on the inclusion and exclusion criteria for this protocol. For subjects who are eligible, the Study Day -5 (Cohort 1) or Study Day -2 (Cohort 2) visit will be scheduled for initiation of JNJ-64281802.

For Cohort 1: Subjects will present to the inpatient unit on Study Day -6. After eligibility criteria have been reviewed and confirmed, subjects will be admitted during this period of intensive PK sampling. Dosing with JNJ-64281802 or placebo will begin on Study Day -5. Discharge will occur on Study Day -4. Dosing with JNJ-64281802 will be observed in-clinic on Days -5, -4, -1, 1, 3, 5, 7, 9, 11, 14, 16, 18, and 21. Subjects will have phone contact on Days -3, -2, 2, 4, 6, 8, 10, 12, 13, 15, 17, 19, and 20 to record time of dose, time of last food intake, and review AEs and concomitant therapy. Daily dosing with JNJ-64281802 or placebo will occur from Study Day -5 through Study Day 21. On Study Day 21 subjects will present to the unit for a second intensive PK sampling period for a full day. On Study Day 1, all subjects will be challenged with rDEN3delta30.

For Cohort 2: Subjects will present to the inpatient unit on Study Day -3. After eligibility criteria have been reviewed and confirmed, subjects will be admitted during this period of intensive PK sampling. Dosing with JNJ-64281802 or placebo will begin on Study Day -2. Discharge will occur on Study Day 1. Dosing with JNJ-64281802 will be observed in-clinic on Days -2, -1, 1, 4, 6, 8, 11, 13, 15, 18, and 21 for the daily dosing regimen and on Days -2, -1, 1, 8 and 15 for the weekly dosing regimens. In the daily dosing regimen with JNJ-64281802 or placebo, twice daily dosing will occur from Study Day -2 to Study Day -1, and daily dosing from Study Day 1 to Study Day 21. In the weekly dosing regimens, twice daily dosing will occur from Study Day -2 to Study Day -1, and weekly dosing which will occur on Study Day 1, Study Day 8, and Study Day 15. On Study Day 21 for the daily regimen, and on Study Day 15 for the weekly regimens, subjects will present to the unit for a second intensive PK sampling period for a full day. On Study Day 1, all subjects will be challenged with rDEN3delta30.

During the inpatient visits on Study Day -6 to -4 (Cohort 1) and Study Day -3 to 1 (Cohort 2), the subjects will be evaluated by a clinician and will have blood drawn for clinical laboratory studies, virologic assays, and immunologic assays. During the outpatient visits subjects will return to the clinic for evaluation and for blood draw as specified in the Schedule of Procedures. Study Day 85 will be the final visit for Cohort 1. Study Day 85 will be the final visit for Cohort 2*. Subjects will have their temperature measured in clinic or measure their temperatures at home twice daily from Study Day 1 through Study Day 29.

ELIGIBILITY:
Inclusion Criteria for receipt of Study Drug:

1. Male or female.
2. 18 to 55 years of age, inclusive, at time of screening.
3. Healthy on the basis of physical examination, medical history, and vital signs performed at screening.
4. Healthy on the basis of clinical laboratory tests performed at screening.
5. Must pass the comprehension assessment indicating that the participant understands the purpose, procedures, and potential risks and benefits of the study, after reading the informed consent and after the investigator or designee has provided detailed information on the study and answered the potential participant's questions.
6. Must have a body mass index between 18.0 and 35.0 kg/m2, inclusive.
7. Must have a normal electrocardiogram (ECG, test which displays a person's heartbeat) at screening.
8. Must have a blood pressure (after lying face up for greater than or equal to 5 minutes) between 90 and 140 mmHg systolic and less than or equal to 90 mmHg diastolic at screening.
9. Must complete the informed consent process independently and without assistance and sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.
10. All persons of childbearing potential must have a negative pregnancy test at screening.
11. A volunteer must be:

    1. Not of childbearing potential, or
    2. Of childbearing potential and practicing a highly effective, preferably user independent method of contraception and agrees to remain on a highly effective method while receiving study drug and until 90 days after the last dose of study drug.
12. A person of childbearing potential must agree not to donate eggs for the purposes of assisted reproduction during the study and for 90 days after the last dose of study drug.
13. During the study and for 90 days after the last dose of study drug, persons who are having sexual relationships in which their partner may become pregnant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. Persons who are having sexual relationships in which their partner may become pregnant should also be advised of the benefit for their partner to use a highly effective method of contraception as condoms may break or leak.
14. A sperm-producing participant must agree not to donate sperm for the purpose of reproduction during the study and for 90 days after the last dose of study drug.
15. Must be willing and able to adhere to the study requirements and lifestyle restrictions:

    * Do not take any restricted medications/treatments
    * Agree to follow all study requirements
    * No unusual strenuous exercise
    * Must not donate blood or blood products within 6 months after last dose of study drug
    * Must not participate in another investigational study during the study or within 90 days after last dose of study drug
    * Must not travel to any dengue-endemic region (as defined by the United States Centers for Disease Control and Prevention
    * Must limit the use of food or drinks/beverages containing alcohol to the absolute minimum from 48 hours before first dose of study drug until Day 85.
    * Must refrain from consumption of grapefruit or grapefruit juice, energy drinks, excessive use of caffeine from 7 days before first dose of study drug until Day 85
    * May not use drugs of abuse (including amphetamine, barbiturate, cocaine, methadone, and opiates) until 3 weeks after the last dose of study drug.
    * Should not consume any food containing poppy seeds or codeine-containing formulation starting 72 hours before the screening visits and before any visit during the follow-up phase (to avoid a false-positive urine drug test).
    * Should follow the instructions for the timing of the standardized meals
16. Available for the duration of the study, which is approximately 85 days after injection of the dengue virus.

Exclusion Criteria for receipt of Study Drug:

1. History of liver or renal impairment; significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, constipation lasting greater than 2 days), endocrine, neurologic, hematologic, rheumatologic, neoplastic, autoimmune, or metabolic disturbances.
2. Known allergies, hypersensitivity, or intolerance to the study drug (JNJ-64281802) or its inactive substances, or an acute, life threatening allergic reaction or swelling following study drug administration.
3. History of a severe allergic reaction or anaphylaxis (which is a severe, potentially life-threatening allergic reaction).
4. Taken any substances or therapies that are not allowed before the first dose of study drug.
5. Received an investigational intervention or participated in another investigational clinical trial (including investigational vaccines) within 6 months before first dose of study drug, or is currently enrolled in an investigational study, or is planning to be enrolled in an investigational study within 90 days after last dose of study drug. With the exception of participation in COVID-19 vaccine trials and receipt COVID-19 vaccines licensed or under Emergency Use Authorization which can be received at any time.
6. Persons of childbearing potential only: Pregnant as determined by a positive pregnancy blood test, breastfeeding, or planning to become pregnant during the study or within 90 days after last dose of study drug.
7. Plans to impregnate and help conceive a child during the study or within 90 days after last dose of study drug.
8. Any condition for which, in the opinion of the study doctor, participation would not be in the best interest of the participant.
9. Blood test confirming current infection with human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2), hepatitis B virus (HBV), or hepatitis C virus (HCV), or blood test confirming past or current infection with any of the following flaviviruses: dengue, Zika virus (ZIKV), West Nile virus, or St. Louis Encephalitis (SLE) virus or vaccination for dengue, Zika virus, or Japanese Encephalitis virus (JEV) Note: Blood laboratory testing will assess the presence of antibodies at screening.
10. Recent (in the past 4 weeks) travel to any dengue-endemic region (as defined by the US CDC) or having definite plans to travel to a dengue endemic region, during the study. Potential participants may be eligible for enrollment greater than or equal to 4 weeks after their return from a dengue-endemic region.
11. Received or plans to receive:

    1. Licensed live attenuated vaccines - within 28 days before first dose of study drug until 28 days after last dose of study drug.
    2. Other licensed (not live) vaccines - within 14 days before first dose of study drug until 14 days after last dose of study drug.
    3. COVID-19 vaccines, either licensed or under EUA, are allowed at any time during the study however every effort will be made to avoid the above windows of time of administration.

    Note: Vaccinations against DENV and Zika virus are not allowed until 90 days after last dose of study drug.
12. Employee of the study doctor or study site with direct involvement in the proposed study or other studies under the direction of that study doctor or study site, as well as family members of the employees or the investigator.
13. Any clinically relevant skin disease in the past 6 months, such as active dermatitis, active eczema, drug rash, psoriasis, and urticaria.
14. Having donated or lost greater than 1 unit of blood (500 mL) within 30 days or greater than 1 unit of plasma (250 mL) within 7 days before first dose of study drug or having the intention to donate blood or blood products during the study and within 6 months after last dose of study drug.
15. Receipt of blood products within the past 6 months of initiation of study drug or anticipated receipt of any blood products during the 28 days following dengue virus injection.
16. Known or suspected congenital or acquired immunodeficiency or use of immunosuppressive corticosteroids (excluding topical and nasal) or immunosuppressive drugs within 28 days before first dose of study drug until 28 days following the last dose of study drug.

    a. An immunosuppressive dose of corticosteroids is defined as greater than or equal to10 mg prednisone equivalent per day for grater than or equal to 14 days.
17. Use of any strong cytochrome P450 (CYP) 3A4 inhibitors (eg, clarithromycin, itraconazole), CYP3A4 inducers (eg, phenytoin, rifampin), or substrates for CYP3A4 (eg, midazolam, triazolam), CYP2C8 (eg, repaglinide), CYP2C9 (eg, warfarin, tolbutamide), BCRP (eg Pravastatin and folic acid), or CYP2C19 (eg, S-mephenytoin, omeprazole) within 14 days before first dose of study drug. Certain other medications are allowed including metformin, levothyroxine, H1 and H2 receptor antagonists, weak CYP3A4 inhibitors, selective serotonin reuptake inhibitors, selective norepinephrine reuptake inhibitors, tricyclic anti-depressants, anxiolytics, and benzodiazepines.
18. Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by participant history, or positive test result(s) for drugs of abuse (including amphetamine, barbiturate, benzodiazepine, cocaine, methadone, and opiates) at screening.
19. Behavioral, cognitive, or psychiatric disease that affects the subject's ability to understand and cooperate with the requirements of the study protocol.
20. Severe asthma (emergency room visit or hospitalization within the last 6 months).
21. Asplenia (the absence of a spleen).
22. Refusal to allow specimen storage for future research.
23. History of risk factors for life-threatening heart rhythm disturbance which includes heart failure, low potassium levels in the blood, family history of fast, chaotic heartbeats known as Long QT Syndrome.

Exclusion Criteria for dengue virus injection:

1. Body temperature greater than or equal to 38.0°C (100.4°F), confirmed by repeat measurements at least 10 minutes after the first measurement.
2. Acute illness.
3. Any other clinical or laboratory finding that would exclude the participant from inoculation (including, but limited to, a positive urine/serum pregnancy test), as assessed by the study doctor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health
Locations (2):
- United States (2):
  - Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland
  - University of Vermont Medical Center (UVMMC), Clinical Research Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durbin AP, Van Wesenbeeck L, Pierce KK, Herrera-Taracena G, Ebone L, Buelens A, Lutton P, Sabundayo BP, Van Eygen V, De Clerck K, Fetter I, Voge NV, Fang X, Goeyvaerts N, Vandendijck Y, Mayfield J, Lenz O, De Meyer S, Kakuda TN, He H, Amaro-Carambot E, Akli RD, Carmolli M, De Marez T, Whitehead SS, Van Loock M, Rasschaert F. Daily Mosnodenvir as Dengue Prophylaxis in a Controlled Human Infection Model. N Engl J Med. 2025 Nov 27;393(21):2107-2118. doi: 10.1056/NEJMoa2500179. PMID 41297006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study follows an adaptive 2-stage design consisting of 2 cohorts enrolled in a staggered manner. Unblinded interim analysis of Cohort 1 was performed to determine the dosing regimens for Cohort 2 and provided results for the primary outcome.
  Cohort 2 was recently unblinded (data analysis is in process) and Cohort 2 is not part of the primary outcome assessment. Therefore, it cannot yet be fully represented in the record (i.e., results).
Groups:
- Cohort 1 - Group 1 JNJ High Dose: JNJ-64281802 (high dose: 600-mg loading dose for 5 days/200-mg maintenance dose for 21 days)
- Cohort 1 - Group 2 JNJ Medium Dose: JNJ-64281802 (medium dose: 200-mg loading dose for 5 days/50-mg maintenance dose for 21 days)
- Cohort 1 - Group 2 JNJ Low Dose: JNJ-64281802 (low dose: 40-mg loading dose for 5 days/10-mg maintenance dose for 21 days)
- Cohort 1 - Group 1/2 Placebo: Placebo (no therapeutic effect). Group 1 Placebo and Group 2 Placebo are combined in one category to be consistent with how data was analyzed. Group 2 placebo were not analyzed on their own (group 1/2 placebos were combined during analysis).
- Cohort 2 - Group 3 JNJ Daily Dose: JNJ-64281802 800mg-BID for 2 days loading dose followed by 250-mg daily maintenance dose for 21 days)
- Cohort 2 - Group 4 JNJ Weekly Dose: JNJ-64281802 450mg-BID for 2 days loading dose followed by 1200-mg weekly maintenance dose for 15 days)
- Cohort 2 - Group 5 JNJ Weekly Dose: JNJ-64281802 250-mg BID for 2 days loading dose followed by 500-mg weekly maintenance dose for 15 days)
- Cohort 2 - Group 3,4,5 Placebo: Placebo (no therapeutic effect). Group 3, 4, 5 Placebo are combined in one category to be consistent with how data will be analyzed.
Period: Overall Study
Arm/Group | Cohort 1 - Group 1 JNJ High Dose | Cohort 1 - Group 2 JNJ Medium Dose | Cohort 1 - Group 2 JNJ Low Dose | Cohort 1 - Group 1/2 Placebo | Cohort 2 - Group 3 JNJ Daily Dose | Cohort 2 - Group 4 JNJ Weekly Dose | Cohort 2 - Group 5 JNJ Weekly Dose | Cohort 2 - Group 3,4,5 Placebo
Started | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6
Completed | 10 | 6 | 6 | 7 | 6 | 7 | 6 | 6
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group 1 Placebo and Group 2 Placebo are combined in one category to be consistent with how data was analyzed. Group 2 placebo were not analyzed on their own (group 1/2 placebos were combined during analysis).
Groups:
- Cohort 1 - Group 1 and Group 2 Placebo: Placebo (no therapeutic effect). Group 1 Placebo and Group 2 Placebo are combined in one category to be consistent with how data was analyzed. Group 2 placebo were not analyzed on their own (group 1/2 placebos were combined during analysis).
- Cohort 2 - Group 3 JNJ Daily Dose: JNJ-64281802 (daily dose: 800-mg BID loading dose for 2 days/250-mg daily maintenance dose for 21 days).
- Cohort 2 - Gorup 4 JNJ Weekly Dose: JNJ-64281802 (weekly dose: 450-mg BID loading dose for 2 days/1200-mg weekly maintenance dose for 15 days).
- Cohort 2 - Group 5 JNJ Weekly Dose: JNJ-64281802 (weekly dose: 250-mg BID loading dose for 2 days/500-mg weekly maintenance dose for 15 days).
- Cohort 2 - Group 3, Group 4 and Group 5 Placebo: Placebo (no therapeutic effect). Group 3 Placebo, Group 4 Placebo and Group 5 Placebo are combined in one category to be consistent with how data will be analyzed.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Group 1 JNJ High Dose | Cohort 1 - Group 2 JNJ Medium Dose | Cohort 1 - Group 2 JNJ Low Dose | Cohort 1 - Group 1 and Group 2 Placebo | Cohort 2 - Group 3 JNJ Daily Dose | Cohort 2 - Gorup 4 JNJ Weekly Dose | Cohort 2 - Group 5 JNJ Weekly Dose | Cohort 2 - Group 3, Group 4 and Group 5 Placebo | Total
Number analyzed (Participants) | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 4 | 4 | 1 | 4 | 4 | 4 | 33
  Male | 4 | 1 | 2 | 4 | 5 | 3 | 2 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 6 | 5 | 7 | 6 | 7 | 6 | 5 | 53
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 3 | 3 | 1 | 2 | 0 | 2 | 19
  White | 3 | 2 | 2 | 3 | 5 | 5 | 5 | 3 | 28
  More than one race | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56
PRNT (50) DENV [Number; unit: participants] — PRNT(50) is defined as the highest dilution of antibody that reduces the number of foci or plaques by 50% compared to the plaque titer of the virus [DENV-1] alone. [Indicator of prior exposure to DENV-1].
  participants
    PRNT (50) DENV-1 <=10 | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56
    PRNT (50) DENV-2 <=10 | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56
    PRNT (50) DENV-3 <=10 | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56
    PRNT (50) DENV-4 <=10 | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6 | 56

OUTCOME MEASURES:

1. Primary Outcome: Assess the Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo in Terms of Reduction of Dengue Infection.
Description: Area under the DENV-3 RNA viral load (VL) concentration-time curves from immediately before inoculation (baseline on Day 1) until Day 29. Cohort 2 was recently unblinded (data analysis is in process) and Cohort 2 is not part of the primary outcome assessment. Therefore, it cannot yet be fully represented in the record (i.e., results).
Time Frame: 28 days
Population: Note group 1 placebo and group 2 placebo are combined per data analysis plan.
Measure: Least Squares Mean (90% Confidence Interval); unit: log10 RNA copies/mL/days
Groups:
- Cohort 1 Group 1 - JNJ High Dose: JNJ-64281802 (high dose: 600-mg loading dose for 5 days/200-mg maintenance dose for 21 days)
- Cohort 1 Group 2 - JNJ Low Dose: JNJ-64281802 (Low dose: 40-mg loading dose for 5 days/10-mg maintenance dose for 21 days)
- Cohort 1 Group 2 - JNJ Medium Dose: JNJ-64281802 (Medium dose: 200-mg loading dose for 5 days/50-mg maintenance dose for 21 days)
- Cohort 1 Group 1/2 Placebo: Placebo (no therapeutic effect)
Arm/Group | Cohort 1 Group 1 - JNJ High Dose | Cohort 1 Group 2 - JNJ Low Dose | Cohort 1 Group 2 - JNJ Medium Dose | Cohort 1 Group 1/2 Placebo
Number analyzed (Participants) | 9 | 6 | 6 | 7
log10 RNA copies/mL/days | 3.00 [2.4 to 3.6] | 5.2 [4.5 to 5.9] | 4.7 [4.0 to 5.4] | 5.0 [4.4 to 5.6]

2. Secondary Outcome: Number of Adverse Events to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Time Frame: 85 Days
Population: Analysis of Cohort 1 data (Groups 1, 2). Note n=29 (not 31) as 2 subjects were excluded from efficacy analysis due to withdrawal prior to DENV-3 inoculation [1 subject randomized to placebo w/d due to SAE; 1 subject randomized to high dose group chose to w/d]. The two subjects who withdrew from the study early are excluded from efficacy analysis but are included in the safety analysis. Also note group 1 placebo and group 2 placebo are combined per sponsor data analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Group 1 Placebo and Cohort 1 Group 2 Placebo: Placebo (no therapeutic effect). Combined Cohort 1 Group 1 Placebo + Cohort 1 Group 2 Placebo.
- Cohort 2 - Group 4 JNJ Weekly Dose: JNJ-64281802 (weekly dose: 450-mg BID loading dose for 2 days/1200-mg weekly maintenance dose for 15 days).
- Cohort 2 - Group 3, Group 4, and Group 5 Placebo: Placebo (no therapeutic effect). Group 3 Placebo, Group 4 Placebo and Group 5 Placebo are combined in one category to be consistent with how data will be analyzed.
Arm/Group | Cohort 1 - Group 1 JNJ High Dose | Cohort 1 - Group 2 JNJ Medium Dose | Cohort 1 - Group 2 JNJ Low Dose | Cohort 1 Group 1 Placebo and Cohort 1 Group 2 Placebo | Cohort 2 - Group 3 JNJ Daily Dose | Cohort 2 - Group 4 JNJ Weekly Dose | Cohort 2 - Group 5 JNJ Weekly Dose | Cohort 2 - Group 3, Group 4, and Group 5 Placebo
Number analyzed (Participants) | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6
Participants
  Participants with 1 or more AE (Any AE) | 11 | 6 | 6 | 8 | 6 | 7 | 6 | 6
  Participants with 1 or more AE related to study treatment | 5 | 4 | 3 | 3 | 1 | 0 | 3 | 2
  Participants with 1 or more AE related to inoculation with DENV-3 | 3 | 5 | 5 | 5 | 0 | 3 | 2 | 4
  Participants with 1 or more AE leading to discontinuation of any study treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Participants with 1 or more AE leading to termination of study participation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Participants with 1 or more AE of Mild severity | 5 | 2 | 2 | 3 | 5 | 5 | 4 | 3
  Participants with 1 or more AE of Moderate severity | 5 | 3 | 4 | 4 | 1 | 0 | 2 | 0
  Participants with 1 or more AE of Severe severity | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 3
  Participants with 1 or more AE of Life-Threatening severity | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Participants with 1 or more serious AE | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Participants with 1 or more serious AE related to study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with 1 or more serious AE related to inoculation with DENV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Physical Examinations to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Time Frame: 99 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Recording of Vital Signs to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Description: Body temperature will be recorded twice daily by study staff and/or by the participants from Day 1 up to and including Day 29; pulse (bpm), systolic and diastolic blood pressure (mmHg) measured on each clinic visit.
Time Frame: 99 weeks
Reporting Status: Not Posted

5. Secondary Outcome: 12-lead ECG With Measurement of QTcF to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Time Frame: 99 weeks
Reporting Status: Not Posted

6. Secondary Outcome: 12-lead ECG With Measurement of QRS Interval to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Time Frame: 99 weeks
Reporting Status: Not Posted

7. Secondary Outcome: 12-lead ECG With Measurement of PR Interval to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Time Frame: 99 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Clinical Laboratory Assessments to Assess the Safety and Tolerability of the Study Drug (JNJ 64281802).
Time Frame: 99 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Assess the Dengue Infection-associated Adverse Events (Unwanted Medical Occurrence).
Description: Occurrence and severity of DENV infection associated AEs.
Time Frame: 99 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo by Reviewing the Area Under the log10-transformed DENV 3 RNA VL Concentration-time Curves From Immediately Before Inoculation (Baseline on Day 1) Until Day 29 (AUCD1 D29 [log10 VL])
Time Frame: 99 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo by Reviewing the Peak of Detectable DENV-3 RNA (log10 VL).
Time Frame: 99 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo for Duration in Days of Detectable DENV-3 RNA.
Time Frame: 99 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo Time to First Onset by Days of Detectable DENV 3 RNA.
Time Frame: 99 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo Based on Presence of Detectable DENV-3 RNA as Measured by PCR (log10 VL) or Culture (log10 VL).
Time Frame: 99 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo on Area Under the Infectious Viremia Curves From Immediately Before Inoculation (Baseline on Day 1) Until Day 29.
Time Frame: 99 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo on the Area Under the log10-transformed Viremia Curves.
Time Frame: 99 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo Peak of Detectable Viremia Level
Time Frame: 99 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo on the Duration of Detectable Viremia.
Time Frame: 99 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo on Time to First Onset of Detectable Viremia.
Time Frame: 99 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Antiviral Activity of the Study Drug (JNJ 64281802) Versus Placebo on Presence of Detectable Viremia.
Time Frame: 99 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Assess How the Body Handles the Study Drug (JNJ-64281802) Following Repeated Oral Dosing. Using Pharmacokinetic Analysis From Repeated Blood Samples Taken at Specified Time Points After Drug Administration During 2 Inpatient Stays.
Description: Blood samples will be taken for measurement of plasma concentrations of JNJ-64281802 at specific time points in the study. Additional PK sampling may be performed on the non-intensive PK days (eg, in the event of an overdose) on other time points, in consultation with the JNJ drug development team.
  Plasma samples will be analyzed to determine concentrations of JNJ-64281802 using a validated, specific, and sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) method under the supervision of the DDT's Bioanalytical Laboratory Department of Bioanalysis.
Time Frame: 99 weeks
Reporting Status: Not Posted

22. Secondary Outcome: Cmax: Maximum Observed Analyte Concentration of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Cmin: Minimum Observed Analyte Concentration of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

24. Secondary Outcome: Ctrough: Observed Analyte Concentration Just Before the Beginning or at the End of a Dosing Interval of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

25. Secondary Outcome: Cavg: Average Analyte Concentration Over the Dosing Interval (τ) Calculated as AUCτ/τ of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

26. Secondary Outcome: Tmax: the Actual Sampling Time to Reach the Maximum Observed Analyte Concentration of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

27. Secondary Outcome: FI: Percentage Fluctuation (Variation) Between Maximum and Minimum Analyte Concentration at Steady-state, Calculated as 100 x ([Cmax - Cmin] / Cavg) of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

28. Secondary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve During the Dosing Interval (t Hours); Calculated by Linear-linear Trapezoidal Summation of JNJ-64281802
Time Frame: 99 weeks
Reporting Status: Not Posted

29. Secondary Outcome: Occurrence and Magnitude of Anti-DENV-3 Total IgM Antibody Titers to Assess the Anti-Dengue Immune Response.
Time Frame: 99 weeks
Reporting Status: Not Posted

30. Secondary Outcome: Occurrence and Magnitude of Anti-DENV-3 Total IgG Antibody Titers to Assess the Anti-Dengue Immune Response.
Time Frame: 99 weeks
Reporting Status: Not Posted

31. Secondary Outcome: Time to First Onset of Anti-DENV-3 Total IgM Antibody Titers to Assess the Anti-Dengue Immune Response.
Time Frame: 99 weeks
Reporting Status: Not Posted

32. Secondary Outcome: Time to First Onset of Anti-DENV-3 Total IgG Antibody Titers to Assess the Anti-Dengue Immune Response.
Time Frame: 99 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data for cohort 1 was collected for the duration of the enrollment period (90 days total) in relation to baseline. Subjects began the study drug (or placebo) on Day -5 followed by challenge with DENV-3 on Day 1, and were followed for AE's through Day 85.
Groups:
- JNJ-64281802 High Dose: JNJ-64281802 High Dose n=11
- Placebo Cohort 1: Placebo Cohort 1 n=8
- JNJ-64281802 Medium Dose: JNJ-64281802 Medium dose n=6
- JNJ-64281802 Low Dose: JNJ-64281802 Low dose n=6
- JNJ-64281802 Daily Dose (Cohort 2 Group 3): JNJ-64281802 Daily Dose (Cohort 2 Group 3) n=6
- JNJ-64281802 Weekly Dose (Cohort 2 Group 4): JNJ-64281802 Weekly Dose (Cohort 2 Group 4) n=7
- JNJ-64281802 Weekly Dose (Cohort 2 Group 5): JNJ-64281802 Weekly Dose (Cohort 2 Group 5) n=6
- Placebo Cohort 2: Placebo Cohort 2 n=6
Arm/Group | JNJ-64281802 High Dose | Placebo Cohort 1 | JNJ-64281802 Medium Dose | JNJ-64281802 Low Dose | JNJ-64281802 Daily Dose (Cohort 2 Group 3) | JNJ-64281802 Weekly Dose (Cohort 2 Group 4) | JNJ-64281802 Weekly Dose (Cohort 2 Group 5) | Placebo Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/8 | 0/6 | 0/6 | 0/6 | 1/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 11/11 | 8/8 | 6/6 | 6/6 | 6/6 | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-64281802 High Dose (N=11) | Placebo Cohort 1 (N=8) | JNJ-64281802 Medium Dose (N=6) | JNJ-64281802 Low Dose (N=6) | JNJ-64281802 Daily Dose (Cohort 2 Group 3) (N=6) | JNJ-64281802 Weekly Dose (Cohort 2 Group 4) (N=7) | JNJ-64281802 Weekly Dose (Cohort 2 Group 5) (N=6) | Placebo Cohort 2 (N=6)
Creatinine Kinase High (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
AST increased (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug overdose (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-64281802 High Dose (N=11) | Placebo Cohort 1 (N=8) | JNJ-64281802 Medium Dose (N=6) | JNJ-64281802 Low Dose (N=6) | JNJ-64281802 Daily Dose (Cohort 2 Group 3) (N=6) | JNJ-64281802 Weekly Dose (Cohort 2 Group 4) (N=7) | JNJ-64281802 Weekly Dose (Cohort 2 Group 5) (N=6) | Placebo Cohort 2 (N=6)
Headache (General disorders) | 6 | 6 | 3 | 6 | 4 | 3 | 3 | 5
Fever (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Dengue-like rash (Infections and infestations) | 3 | 7 | 4 | 5 | 1 | 1 | 1 | 4
Local Tenderness (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Elevated ALT (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Infections and infestations) | 0 | 3 | 3 | 5 | 1 | 2 | 0 | 4
Arthalgia (Infections and infestations) | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 1
Retroorbital Pain (Infections and infestations) | 0 | 3 | 2 | 3 | 3 | 0 | 0 | 3
Fatigue (Infections and infestations) | 3 | 5 | 1 | 4 | 2 | 3 | 3 | 5
Nausea (Infections and infestations) | 4 | 4 | 1 | 4 | 1 | 2 | 2 | 2
Prolonged PT (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Prolonged PTT (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Increased Cholesterol (Investigations) | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Elevated lipase (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT05048875/Prot_SAP_000.pdf